CLINICAL TRIAL: NCT04760886
Title: Comparing Paediatric Trauma Presentations in a Rural District General Hospital and an Urban Major Trauma Centre: a Retrospective Cohort Study
Brief Title: Paediatric Rural vs Urban Trauma
Status: Completed | Type: Observational
Sponsor: Mrs Jennifer M Dunn (Other)
Responsible Party: Sponsor-Investigator, Mrs Jennifer M Dunn, ST3 (Trauma and Orthopaedics), NHS Highland
Organization: NHS Highland (Other)
Other Study IDs: Paediatric trauma study
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Paediatric Trauma
Keywords: Paediatric trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urban trauma cohort: All paediatric trauma admissions in an urban, MTC treated operatively, isolated from a departmental trauma list between 1st April 2019- 1st April 2021
  Interventions: Other: Type of hospital (rural DGH vs Urban MTC)
- Rural trauma cohort: All paediatric trauma admissions in a rural district general, treated operatively, isolated from a departmental trauma list between 1st April 2019- 1st April 2021
  Interventions: Other: Type of hospital (rural DGH vs Urban MTC)

INTERVENTIONS:
Other: Type of hospital (rural DGH vs Urban MTC) — In this small cohort study, the hospital in which the patients were treated was the intervention. One was in a rural area and was a district general, whereas one was in an urban enviroment and was a major trauma centre.

SUMMARY:
Retrospective cohort study examining paediatric trauma admission over 1 year in a rural hospital vs urban centre

DETAILED DESCRIPTION:
As above. All patient data was anonymised.

ELIGIBILITY:
Inclusion Criteria:

* All paediatric trauma in each centre over the above time frame, treated operatively, seen on an acute orthopaedic take

Exclusion Criteria:

* Adults, non-operative trauma

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: age 0-16yr olds with paediatric trauma, treated operatively.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Type of operation performed | 1st April 2019- 1st April 2020
  Type of orthopaedic intervention documented
Distribution of type of paediatric trauma | 1st April 2019- 1st April2020
  Sub-types of fractures seen documented

SECONDARY OUTCOMES:
Seasonality of trauma | 1st April 2019- 1st April 2020
  winter vs summer months trauma numbers documented

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dunn, Principal Investigator — NHS Highland
Locations (1):
- Jennifer Dunn, Raigmore hospital orthopaedic department, Inverness, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No